CLINICAL TRIAL: NCT07197996
Title: MonitoRing the Effect of Intermittent Pneumatic Compression and TRAnscutaneous Functional electrIcal Stimulation of the Common Peroneal Nerve Using the Geko® Device on Cerebral Haemodynamics in Patients With Ischaemic Strokes (The RETRAIN Trial Phase 2)
Brief Title: The RETRAIN Trial Phase 2
Acronym: RETRAIN 2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firstkind Ltd (Industry)
Collaborators: Innovate UK (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISS-BBF-002; 10038715 (Other Grant/Funding Number: Innovate UK)
Record Dates: First submitted 2025-09-25; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-03

CONDITIONS: Ischaemic Stroke
Keywords: Acute ischemic stroke; Neuromuscular electrostimulation; Effects on cerebral blood flow; Randomised controlled trial; Cerebral blood flow measurements; Stroke rehabilitation
MeSH Terms: conditions — Ischemic Stroke | interventions — Intermittent Pneumatic Compression Devices

STUDY DESIGN:
Intervention Model Description: Randomized, Parallel Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - IPC device (Experimental): IPC sleeves applied bilaterally according to manufacturer's instructions for standard VTE prophylaxis following ischaemic stroke.
  Interventions: Device: Intermittent Pneumatic Compression
- Group 2 - geko® device (Experimental): The geko® device is a disposable, battery-powered neuromuscular electrostimulation device applied bilaterally to the peroneal nerve at the knee. It delivers low-frequency stimulation to activate the calf and foot muscle pumps, enhancing venous return and microcirculatory blood flow. Devices will be applied according to the manufacturer's instructions for VTE prophylaxis.
  Interventions: Device: geko® T3

INTERVENTIONS:
Device: Intermittent Pneumatic Compression — The IPC arm will use the Kendall SCD™ 700 Sequential Compression System, a routinely employed device for VTE prophylaxis in stroke patients. In this study, IPC sleeves will be applied bilaterally to the legs within 36 hours of stroke onset and operated according to the manufacturer's instructions. The intervention is distinguished by its cyclical external leg compression to enhance venous return, and it serves as the comparator to the geko® device for evaluating effects on cerebral blood flow and haemodynamics.
  Other Names: Kendall SCD™ 700 Sequential Compression System
  Arms: Group 1 - IPC device
Device: geko® T3 — The geko® T3 device is a small, disposable, battery-powered neuromuscular electrostimulation device manufactured by Firstkind Ltd. In this study, the geko® will be applied bilaterally to the common peroneal nerve at the knee within 36 hours of stroke onset. It delivers transcutaneous electrical stimulation at 1 Hz, producing involuntary rhythmic foot dorsiflexion to activate the calf and foot muscle pumps. The intervention is distinguished from IPC by its mechanism of action (neuromuscular stimulation vs. external compression) and will be evaluated for its impact on cerebral haemodynamics, neurovascular coupling, and dynamic cerebral autoregulation during VTE prophylaxis.
  Other Names: geko® device, neuromuscular electrostimulation
  Arms: Group 2 - geko® device

SUMMARY:
Ischaemic strokes, caused by a disruption in the brain's blood supply, are the second leading cause of death and disability in the United Kingdom. This single-center prospective randomised study aims to measure cerebral blood flow and oxygen delivery in patients who have recently suffered an ischaemic stroke and are using either the geko® neuromuscular electrostimulation device or an intermittent pneumatic compression (IPC) device as part of their routine clinical care.

The geko® device stimulates a nerve in the lower leg, inducing muscle contractions that enhance blood circulation. The IPC device applies controlled external pressure through compressed air and a pump, cyclically inflating and deflating chambers in a sleeve worn on the leg. This mimics the action of calf muscles to promote blood flow.

The primary objective of this study is to assess the effect of the geko® and IPC devices on cerebral blood flow in stroke patients, specifically during the hyperacute phase (within 36 hours) following an ischaemic stroke. Both devices will be used as part of standard care for VTE prevention. Cerebral blood flow will be measured using functional near-infrared spectroscopy (fNIRS) and electroencephalography (EEG).

DETAILED DESCRIPTION:
This study is a randomised trial at a single centre, comparing brain blood flow and activity patterns when two standard treatments for preventing blood clots (VTE) are used following a stroke.

Who Can Take Part?

Patients will be identified for the study as part of their routine hospital care when they arrive at hospital through the emergency department. To take part they must:

1. Be 18 years or older
2. Have had an ischaemic stroke confirmed by a stroke doctor
3. Be within 36 hours of stroke symptom onset
4. Be unable to stand or move around
5. Have had a CT or MRI scan confirming no bleeding in the brain

What Will Happen?

After confirming eligibility and once consent is given, 80 participants will be randomly assigned to one of two groups during the study period:

Group 1 - IPC device Group 2 - geko® device

Both devices are standard treatments for preventing blood clots.

Study Assessments

Brain blood flow will be measured while participants are sitting upright in bed. Each session will include:

5 minutes with the device switched off 5 minutes with the device switched on

These assessments will take place twice a day for two days (a total of 40 minutes) with a pre-assessment preparation (a total of 80 minutes over the two days). Blood pressure, ECG, temperature, and oxygen levels will be continuously monitored. No follow-up is required after the study.

ELIGIBILITY:
Inclusion Criteria:

1. Adult over 18
2. Patient with ischaemic stroke diagnosis confirmed by a stroke physician.
3. Within 36 hours of symptom onset.
4. Unable to stand or mobilise without assistance.
5. No intracerebral haemorrhage as ruled out by computerised tomography (CT) or Magnetic Resonance Imaging (MRI) scan.

Exclusion Criteria:

1. Inability to gain consent from the patient, or a declaration from a Personal Consultee or Nominated Consultee.
2. Absence of a transient ischaemic attack (TIA).
3. Clinically apparent deep vein thrombosis at screening
4. Patient is expected to require palliative care within 14 days
5. No response to the geko® device i.e. no involuntary rhythmic upward and outward movement of the foot (dorsiflexion) at the maximum tolerable device setting.
6. Contraindications for the use of the geko™ device

   * Allergy to hydrogel constituents
7. Contraindications to IPC

   * Severe peripheral vascular disease
   * Large leg ulcers requiring extensive bandaging (small ulcers or skin breaks with flat coverings are not an exclusion)
   * Severe oedema
   * Leg deformities making appropriate fitting impossible
   * Symptomatic congestive cardiac failure of NYHA class IV (symptoms of heart failure at rest, any physical activity causing further discomfort).
8. Single or double leg amputations.
9. Participation in any other clinical trial
10. Patients must not have a current coronavirus (COVID-19) infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-07-01 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
Change in Cerebral Blood Flow During Device Use | Day 1-2 (within 36 hours of stroke onset; measurements taken twice daily for 2 consecutive days)
  Cerebral blood flow (CBF) will be assessed using functional near-infrared spectroscopy (fNIRS) combined with EEG, beat-to-beat blood pressure, and transcutaneous CO₂ monitoring. Measurements will compare baseline (no device) to during active use of either the Intermittent Pneumatic Compression (IPC) device or the geko® T3 device. The primary analysis will evaluate differences in cerebral haemodynamics between the two randomized intervention groups.

SECONDARY OUTCOMES:
Change in Neurovascular Coupling During Device Use | Day 1-2 (twice daily assessments for 2 consecutive days)
  Changes in neurovascular coupling will be assessed using combined functional near-infrared spectroscopy (fNIRS) and EEG during resting state and during active use of the Intermittent Pneumatic Compression (IPC) device or the geko® T3 device.
Change in Dynamic Cortical Connectivity During Device Use | Day 1-2 (twice daily assessments for 2 consecutive days)
  Functional connectivity between cortical regions will be measured using fNIRS+EEG data during intervention (IPC or geko® device) compared to baseline.
Incidence of Adverse Events | Up to 2 days from enrolment
  Number and type of adverse events observed in participants during and after use of either device.
Incidence of Serious Adverse Events | Up to 2 days from enrolment
  Frequency of serious adverse events, including death, life-threatening illness, permanent impairment, or prolonged hospitalisation
Incidence of Adverse Device Effects | Up to 2 days from enrolment
  Frequency of device-related adverse events such as discomfort, skin irritation, or unexpected physiological responses to device use.
Incidence of Serious Adverse Device Effects | Up to 2 days from enrolment
  Frequency of serious device-related adverse events meeting criteria for seriousness under ISO 14155:2020.
Incidence of Device Deficiencies | Up to 2 days from enrolment
  Frequency and type of device deficiencies (malfunctions, usability issues, or inadequacy of instructions for use) observed during the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Kausik Chatterjee, Study Director — COUNTESS OF CHESTER HOSPITAL NHS FOUNDATION TRUST
Locations (1):
- Countess of Chester Hospital, Chester, Cheshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) underlying the results of this trial (including baseline characteristics, outcome measures, and safety data) will be made available to other researchers upon reasonable request, following publication of the main trial results. Data will be shared through a controlled access process after approval of a research proposal and data sharing agreement. Supporting documents (such as the study protocol and statistical analysis plan) will also be available.
Supporting Information: Study Protocol, SAP
Time Frame: De-identified IPD will be available beginning 12 months after publication of the primary results and for a period of up to 5 years thereafter.
Access Criteria: Researchers must submit a methodologically sound proposal, which will be reviewed by the sponsor and chief investigator. Access will be granted only after a data sharing agreement is signed.